CLINICAL TRIAL: NCT01509274
Title: Treatment of Plantar Fasciitis With Injection af Platelet-rich Plasma Into the Origin of the Plantar Fascia - a Prospective, Randomized and Double Blinded Study.
Brief Title: Treatment of Plantar Fasciitis With Injection af Platelet-rich Plasma Into the Origin of the Plantar Fascia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Bjørn Nedergaard, Cand. Med., Kolding Sygehus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS6000
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Plantar Fasciitis
Keywords: Plantar fasciitis; Plasma; PRP; Heel pain
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Sodium Chloride; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plasma (Experimental)
  Interventions: Biological: Plasma
- Saline (Sham Comparator)
  Interventions: Biological: Saline
- Physiotherapy + heel cap (Active Comparator)
  Interventions: Other: Physiotherapy + heel cap

INTERVENTIONS:
Biological: Plasma — 3 ml plasma injected once into the plantar fascia
  Arms: Plasma
Biological: Saline — 3 ml of saline injected once into the plantar fascia
  Arms: Saline
Other: Physiotherapy + heel cap — Physiotherapy three times a day for 8 weeks. Heel caps until symptoms are gone
  Arms: Physiotherapy + heel cap

SUMMARY:
The purpose of our study is to determine whether one injection with plasma into the origin of the plantar fascia is an effective treatment of plantar fasciitis.

90 patients will be randomized into three groups. 30 patients will be treated with one plasma injection, 30 patients will be treated with one injection with saline and 30 patients will do physiotherapy and use heel cups. The two groups who receive injections will do the same physiotherapy and use heel cups, as the conservatively treated group.

Both groups randomized to receive an injection will have a 10 ml blood sample taken from their cubital vein. The sample is centrifuged for 5 minutes at 5000 rpm. No additives are added. 3 ml of plasma i obtained, and the syringe i blinded. Is the patient randomized to receive an injection with saline, a similar syringe is blinded with 3 ml of saline. The injection into to the origin of the plantar fascia i done 10 minutes after the sample of blood is obtained. The content of the syringe i blinded to both the investigator and the patient.

The injection i performed from the medial aspect of the heel under guidance of ultrasound. No local/systemic analgetic is used. The content of the syringe is spread using peppering technique into the origin of the plantar fascia.

Patients will do questionnaires at inclusion and after 1, 2, 3, 6 and 12 months. The questionaires will be Foot Function Index and SF-36 as well as questions about their use of analgetics, use of heel cups and intensity of their physiotherapy

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 of age
* Sore at the insertion of the plantar fascia on calcaneus
* A VAS score of at least 4 at the insertion of the plantar fascia on calcaneus taking the first step in the morning
* Symptoms for 6 to 12 months
* Ability to understand danish and give informed consent

Exclusion Criteria:

* Previously operated in the same ankle or foot
* Pain anywhere else in the foot on palpation otherwise than at the insertion of the plantar fascia on calcaneus
* Inflammatory disease
* Diabetes
* Formerly rupture of the Achilles tendon
* Formerly treated with plasma injections
* Ongoing infection treated with antibiotics
* Treated with steroid during the trial
* Treatment of the plantar fasciitis exceeding conservative treatment
* Use of crutches, walker or similar
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Pain on a VAS score

SECONDARY OUTCOMES:
Disability

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Nedergaard, Cand. Med., Principal Investigator — Kolding Sygehus
Locations (1):
- Sygehus Lillebælt - Kolding Sygehus, Kolding, Denmark